CLINICAL TRIAL: NCT05382208
Title: Doxycycline for Emphysema in People Living With HIV (The DEPTH Trial)
Acronym: DEPTH
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); University of California, Los Angeles (Other); University of Iowa (Other); University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-02-307/22-04024723; DEPTH-001 (Other: Weill Cornell Medicine); UH3HL154944 (NIH)
Record Dates: First submitted 2022-05-16; First posted 2022-05-19 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Emphysema; HIV
MeSH Terms: conditions — Emphysema | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participant and site personnel will not know which study treatment the participant is receiving.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Doxycycline (Experimental): Doxycycline 100mg orally twice a day
  Interventions: Drug: Doxycycline
- Placebo (Placebo Comparator): Matching placebo orally twice a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Doxycycline — Doxycycline 100 mg orally twice a day.
  Arms: Doxycycline
Drug: Placebo — Matching placebo orally twice a day.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if doxycycline will reduce progression of emphysema in people living with HIV.

The secondary objectives are to examine the effects of doxycycline on change in quantity of emphysema, six minute walk distance, patient reported outcomes, ratio of forced expiratory volume in 1 second and forced vital capacity. Secondary objectives will also describe the safety and tolerability of doxycycline and determine if doxycycline is associated with development of antibiotic-resistant bacterial infections.

DETAILED DESCRIPTION:
This study is a phase II, multicenter, randomized, double-blinded, placebo-controlled clinical trial in approximately 250 people living with HIV who have emphysema.

Eligible participants will be randomized in a 1:1 fashion to doxycycline or placebo. Participants will receive 100 mg doxycycline orally or matched placebo twice a day for 72 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 30 years and older at screening visit.
* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to the enrollment visit, and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load.
* Current or former smoker with at least a 3 pack-year history of cigarette smoking at screening visit.
* Evidence of emphysema on high resolution CT (HRCT) of the chest done at pre-entry visit (Visit 2). Emphysema is defined as either:

  1. Mild, moderate, or severe emphysema assessed by central reader(s) at the CT Imaging Core; or
  2. Quantification of ≥ 5% of voxels with density < -950 Hounsfield Units (HU) as quantified by the CT Imaging Core.

All participants with emphysema by either or both criteria must have ≤ 35% of voxels with density < -950 HU.

* Screening and Entry DLCO measurements must be within 15% of each other. The PFT quality at both visits must be acceptable based on ATS Quality Criteria.

  1. Screening (Visit 1) Pulmonary Function Test meets ATS quality criteria as determined by a central reviewer at the PFT Reading Core (UCLA)
  2. Baseline (Visit 2) Pulmonary Function Test meets ATS quality criteria as determined by the central reviewer at the PFT Reading Core (UCLA), Site Investigator, or DEPTH Trial Leadership.
* HIV-1 RNA level < 200 copies/ml within 90 days prior to the Entry/Baseline visit by any US laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent.
* CD4 cell count > 100 cells/mm3 within 90 days prior to the Entry/Baseline visit.by any US laboratory that has a CLIA certification or its equivalent.
* Stable antiretroviral therapy for greater than or equal to 8 weeks prior to the Entry/Baseline visit. Substitutions of one formulation of a drug for another are not considered changes in antiretroviral therapy for the purpose of defining stable therapy..
* Serum ALT and AST < 3 x upper limit of normal within 60 days prior to the Entry/Baseline visit.
* Participants on therapy for COPD must be on stable therapy for at least 4 weeks prior to the Entry/Baseline visit.
* Documentation of serum alpha-1-antitrypsin level above the lower limit of normal from a test done at any time prior to the Entry/Baseline visit.
* Provision of signed and dated written informed consent.
* Stated willingness to adhere to all study procedures and anticipated availability for the duration of the study.
* Life expectancy > 2 years in the opinion of the site investigator.
* Ability to take oral medication and willingness to adhere to the study drug.
* For individuals of reproductive potential, negative serum or urine pregnancy test with a sensitivity of less than or equal to 25 mIU/mL at the screening visit. This will be repeated at the Entry/Baseline visit.

Exclusion Criteria:

* Pulmonary infection, acute COPD exacerbation, acute opportunistic infection within 30 days prior to the Screening Visit 1 or Entry/Baseline Visit 2.
* Any acute or serious illness requiring systemic treatment and/or hospitalization within 30 days prior to the Entry/Baseline visit.
* Decompensated cirrhosis defined as an acute deterioration in liver function in a patient with cirrhosis and is characterized by jaundice, ascites, hepatic encephalopathy, hepatorenal syndrome or variceal hemorrhage.
* History of, or planned, wedge resection, lobectomy, pneumonectomy, or lung volume reduction surgery.
* History of, or planned, endobronchial valve placement for lung volume reduction.
* Significant parenchymal lung disease other than emphysema or chronic bronchitis (e.g. sarcoidosis, MAI infection, pulmonary fibrosis, lung cancer, bullae/cysts from prior Pneumocystis pneumonia) that would preclude accurate quantification of emphysema.
* Previous allergy or intolerance to doxycycline or other drugs in the tetracycline class (e.g. minocycline, tetracycline).
* Breastfeeding individuals.
* Receipt of any investigational* drug within 30 days prior to the Entry/Baseline visit. Note: for the purpose of this protocol, investigational drug refers to a drug that is not FDA approved for any indication. COVID vaccines available under emergency use authorization are allowed.
* Need for concomitant use of barbiturates; carbamazepine; phenytoin
* Use of systemic retinoids (eg. Isotretinoin [Accutane]) or Vitamin A within 30 days prior to the Entry/Baseline visit. Note: Multivitamin containing Vitamin A use is permitted.
* Use of any systemic antibiotic (e.g., doxycycline or other tetracycline, azithromycin) within 7 days prior to the Entry/Baseline visit.
* Any condition including active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* History of recurrent C. difficile infection or C. difficile infection within 30 days prior to the Entry/Baseline visit.
* Inability to stop supplemental oxygen for 15 minutes to perform a DLCO maneuver.
* Has changes to the chest that preclude adequate HRCT imaging (e.g. Metallic objects in the chest such as shrapnel or pacemaker leads)
* Current receipt of, or anticipated need to initiate, hemodialysis or peritoneal dialysis.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2022-08-22 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Rate of decline (slope) of percent predicted diffusing capacity for carbon monoxide (DLCO) corrected for hemoglobin, carboxyhemoglobin and barometric pressure (indicated as ppDLCOadj) over the 72 week treatment period. | 72 weeks

SECONDARY OUTCOMES:
Change from baseline to week 48 in 6 minute walk test distance. | 48 weeks
Change from baseline to week 72 in 6 minute walk test distance. | 72 weeks
Change from baseline to week 48 in percent predicted diffusing capacity for carbon monoxide (DLCO) corrected for hemoglobin, carboxyhemoglobin and barometric pressure (ppDLCOadj). | 48 weeks
Change from baseline to week 72 in percent predicted diffusing capacity for carbon monoxide (DLCO) corrected for hemoglobin, carboxyhemoglobin and barometric pressure (ppDLCOadj). | 72 weeks
Change from baseline to week 72 in percentage of voxels < -950 Hounsfield Units (HU) | 72 weeks
Change from baseline to week 48 in the COPD Activity Test (CAT) score | 48 weeks
  The COPD Assessment Test (CAT): CAT is an 8-item self-administered questionnaire. Scores range from 0 to 40. Higher scores denote a more severe impact of COPD on a patient's life.
Change from baseline to week 72 in the COPD Activity Test (CAT) score | 72 weeks
  The COPD Assessment Test (CAT): CAT is an 8-item self-administered questionnaire. Scores range from 0 to 40. Higher scores denote a more severe impact of COPD on a patient's life.
Change from baseline to week 48 in St. George's Respiratory Questionnaire (SGRQ) score | 48 weeks
  St. George's Respiratory Questionnaire (SGRQ): SGRQ is a 50-item respiratory disease-specific health-related quality of life (HRQOL) instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Scores range from 0 to 100, with higher scores indicating more limitations.
Change from baseline to week 72 in St. George's Respiratory Questionnaire (SGRQ) score | 72 weeks
  St. George's Respiratory Questionnaire (SGRQ): SGRQ is a 50-item respiratory disease-specific health-related quality of life (HRQOL) instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Scores range from 0 to 100, with higher scores indicating more limitations.
Change from baseline to week 48 in forced expiratory volume in 1 second (FEV1) (L) | 48 weeks
Change from baseline to week 72 in forced expiratory volume in 1 second (FEV1) (L) | 72 weeks
Change from baseline to week 48 in the ratio of forced expiratory volume in 1 second and forced vital capacity (FEV1/FVC) | 48 weeks
Change from baseline to week 72 in the ratio of forced expiratory volume in 1 second and forced vital capacity (FEV1/FVC) | 72 weeks
The number of adverse events | 72 weeks
  The number of adverse events regardless of relatedness to the intervention
The proportion of participants with at least 1 adverse event | 72 weeks
  The proportion of participants with at least 1 adverse event regardless of relatedness to the intervention
The number of serious adverse events. | 72 weeks
  Serious adverse events (SAEs) will include all treatment-emergent SAEs.
The proportion of participants with at least 1 serious adverse event. | 72 weeks
  The proportion of participants with at least 1 Serious adverse event (SAE). SAEs will include all treatment-emergent SAEs.
The proportion of participants with deaths. | 72 weeks
The number of participants permanently discontinuing study medication due to adverse events. | 72 weeks
  The number of participants permanently discontinuing study medication due to treatment-emergent adverse events.
The proportion of participants permanently discontinuing study medication due to adverse events. | 72 weeks
  The proportion of participants permanently discontinuing study medication due to treatment-emergent adverse events.
The number of participants with development of culture proven antibiotic-resistant bacterial infection with reduced susceptibility or resistance to doxycycline (adverse event of special interest). | 72 weeks
The proportion of participants with development of culture proven antibiotic-resistant bacterial infection with reduced susceptibility or resistance to doxycycline (adverse event of special interest). | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marshall J Glesby, MD, PhD, Principal Investigator — Weill Medical College of Cornell University; Cathie Spino, ScD, Principal Investigator — University of Michigan; Robert J Kaner, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (20):
- United States (20):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California Los Angeles, Los Angeles, California
  - University of California San Diego, San Diego, California
  - Miami University, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Tulane University, New Orleans, Louisiana
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - SUNY Downstate Medical School, Brooklyn, New York
  - Weill Cornell Medicine, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University School of Medicine, Durham, North Carolina
  - University of Cincinnati College of Medicine, Cincinnati, Ohio
  - Case Western University, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Temple University, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas, McGovern Medical School, Houston, Texas
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
The de-identified analytic data will be prepared as SAS transport files or ASCII comma-delimited files with accompanying codebooks that describe the data and data structure. The redaction will employ best practices and will be consistent with NHLBI data sharing policies.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study data will be shared through the NHLBI data repository, no later than 3 years after the end of the study or 2 years after the main paper reporting the results of the trial, whichever comes first.
Access Criteria: Data will be shared through the NHLBI Biologic Specimen and Data Repository Information Coordinating Center (BioLINCC).
URL: https://biolincc.nhlbi.nih.gov/home/